CLINICAL TRIAL: NCT03614091
Title: Analgesic and Pulmonary Function Effects of Erector Spinae Plane Block Versus Paravertebral Plane Block for Women's Undergoing Modified Radical Mastectomy; Randomized Comparative Study
Brief Title: Paravertebral Block Versus Erector Spinae Plane Block for Modified Radical Mastectomy in Womens.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, jehan ahmed sayed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AssiutU748918
Record Dates: First submitted 2018-07-13; First posted 2018-08-03 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Pain, Postoperative; Pulmonary Atelectasis; Mastectomy
Keywords: Paravertebral block; Erector spinae plane block; Modified radical mastectomy; respirometer
MeSH Terms: conditions — Pain, Postoperative; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Double Blind (caregiver,outcome Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Paravertebral plane block group (Active Comparator): The TPVB will be administered at the T4 level with the patient in the sitting position.The ultrasound probe will be placed 5 cm from the midline in the craniocaudal direction and moved medially to identify the transverse process and parietal pleura. The superior costotransverse ligament was identified as a collection of homogeneous linear echogenic bands alternating with echo-poor areas running from one transverse process to the next. Bubivacaine0.5%, 20 ml will be deposited in the space between the pleura and the costotransverse ligament.
  Interventions: Procedure: Paravertebral plane block
- Erector spinae plane block group (Active Comparator): the transducer will be placed in a transverse orientation at T5 to T6 to identify the spinous process, lamina, and transverse process .The tip of the transverse process will be centered on the ultrasound screen, and the transducer will be rotated 90 degrees into a longitudinal orientation to obtain a parasagittal view. Depending on the level imaged, 2 or 3 hypoechoic muscle layers were identiﬁed overlying the tip of the transverse processes. From T1 to T5 the erector spinae, rhomboid major and trapezius muscles are visible posterior and superficial to the transverse processes. An 8cm 22-gauge block needle will be Inserted in-plane to the ultrasound beam in a cephalad-to-caudal Direction to place the needle tip between the posterior fascia of Erector spinae and the tip of the targeted transverse process. Following which a total of 20 mL of 0.5%bupivacaine will be injected.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — 20 ml Bupivacaine 0.5% below erector spinae muscle groups
  Other Names: ultrasound guided Erector spinae plane block
  Arms: Erector spinae plane block group
Procedure: Paravertebral plane block — 20 ml Bupivacaine 0.5% between pleura and costotransverse ligament
  Other Names: ultrasound guided thoracic Paravertebral plane block
  Arms: Paravertebral plane block group

SUMMARY:
postoperative pain following Modified radical mastectomy is severe specially after dissection of tissues .paravertebral plane block provides an excellent postoperative analgesia for women's,but it carry the risk of pneumothorax which it reported in some cases.Erector spinae plane block is a recent block has been mentioned in many case reports as a safe,quick and can be used in outpatient setting. we use a comparative study to compare the postoperative analgesia between both blocks and the affection of postoperative pain following both blocks if any on pulmonary functions.

DETAILED DESCRIPTION:
Postoperative pain is one of the commonest problems encountered by anesthesiologists in their practice, especially after radical mastectomy surgeries , in which post-operative pain would cause a restrictive respiratory dysfunction, which is associated with poor postoperative outcomes.

Postoperative pulmonary complications (PPCs) are the leading cause of death and increase hospital care expenditures in cardiothoracic and non- cardiothoracic surgery. Included under the heading of (PPCs) are respiratory failure, pneumonia, atelectasis, and exacerbation of chronic obstructive pulmonary disease.

Modiﬁed radical mastectomy, usually performed for the treatment of breast cancer, is associated with considerable acute postoperative pain and restricted shoulder mobility An estimated 40% of women report significant pain symptoms following mastectomy Poor pain relief has been associated with additional healthcare costs, resource utilization and prolonged inpatient stay after surgery.

the thoracic paravertebral block (TPVB) is the most widely used technique to provide postoperative analgesia after breast surgeries Advantages of a TPVB technique include reduced postoperative pain, analgesic consumption and shorter post anesthesia care unit (PACU) stay There is also evidence to suggest that TPVB may have a favorable impact on cancer recurrence after mastectomy. Paravertebral blockade results in somatosensory and sympathetic blockade after injection of local anesthetic solution to the paravertebral space posterior to the pleura.

Erector spinae plane (ESP) block is a recently described technique which may be an alternative to PVB for providing thoracic analgesia. Numerous case reports and case series describe ESP block for the management of acute and chronic thoracic pain. It involves injection of local anesthetic into the fascial plane deep to erector spinae muscle.

Radiological imaging in a cadaver model has demonstrated that a single injection at the level of the T5 transverse process produced cranio-caudal spread between C7 and T8 . This accounts for the extensive sensory block that has been observed in case reports and is at least as extensive as the spread seen with TPVB ESP is a more superficial block with a better defined end-point - injection between the bony transverse process and erector spinae muscle. A more superficial ultrasound-guided block will be faster to perform and less painful for the patient. Furthermore, ESP does not have the same risk of pneumothorax as TPVB. There have been no randomized controlled trials involving ESP to date. All descriptions of the technique have been in case report / series format.

The investigators hypothesize that ESP block efficacy is not inferior to TPVB with reference to dermatomal sensory spread and analgesic efficacy, while being easier to perform, has less associated discomfort and fewer complication risk ESP has been no randomized in many case trials and they found that it effective as postoperative analgesia in modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade II-III.
* female patients in the age group of 18-50 yr.
* undergoing modiﬁed radical mastectomy under general anesthesia.
* BMI <40 kg.m2.

Exclusion Criteria:

* pre-existing infection at the block site.
* Coagulopathy.
* morbid obesity (BMI >40 kg m-2).
* allergy to local anesthetics.
* decreased pulmonary reserve.
* major cardiac disorders.
* renal dysfunction.
* pre-existing neurological deﬁcits.
* psychiatric illness.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — After providing written informed consent, 40 patients, (American Society of Anesthesia):ASA grade II-III, female patients in the age group of 18-50 yr, who will be undergoing modiﬁed radical mastectomy under general anesthesia will be included
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Tests(PFT) | preoperative and 24 hours postoperative
  Pulmonary function test (PFTs) will be performed for all of them in the day before operation .pulmonary function tests will assess via a portable spirometer (Enraf-Nonius, Model SPIRO 601 Medical Technologies) with the patient in the sitting or semi-recumbent position. PFTs will obtain with the elimination of outliers from data analysis

SECONDARY OUTCOMES:
Opioid consumption | 24 hours postoperatively
  the total dose of nalbuphine in 24 hours
Hospital stay | 72 hours
  postoperative Hospital stay in hours
Dermatomal distribution | 30 minutes after block will be assessed every 5 minutes
  Dermatomal distribution of each block 30 minutes before the surgery (sensory loss tested by pin prick and Autonomic assessment by ethanol alcohol).
Incidence of Side effects and complication during study | 24 hours
  Any side effects or complication will be observed and managed in the first 24 hours postoperative Hours will be recorded: nausea, vomiting, lower limb weakness, Respiratory depression (Decrease in SPo2 of less than 90% Requiring supplementary oxygen), urinary retention, rash and Pruritus will be noted and managed.
Time to first analgesic requirement | 24 hours postoperative
  the time from end of surgery to the first requirement of Postoperative analgesia by measuring verbal numeric rating scale, which will be assessed in 0-0.5-1-2-4-6-8-12-24 hours,Patients will be administered 6mg nalbuphine as rescue analgesia whenever the pain score (VNRS) reached 4 or more.

CONTACTS AND LOCATIONS:
Overall Officials: jehan ahmed sayed, MD, Study Director — Assisstant professor in Anaesthesia and ICU department,faculty of medicine,Assiut University ,egypt; mahmoud abdel aziz ali, PHD, Study Chair — Professor of Anesthesia & ICU Faculty of Medicine - Assiut University,egypt; mahmoud bahaa mousa, M.B.B.Ch, Principal Investigator — assisstant lecturer of Anaesthesia and ICU department,faculty of medicine ,Assiut University,egypt
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayed JA, Hamed R, Abdelraouf AM, El-Hagagy NYM, El Dean Mousa MB, Abdel-Wahab AH. A comparative study of respiratory effects of erector spinae plane block versus paravertebral plane block for women undergoing modified radical mastectomy. BMC Anesthesiol. 2024 Jul 30;24(1):262. doi: 10.1186/s12871-024-02632-4. PMID 39080545